CLINICAL TRIAL: NCT04384250
Title: Genetic Factors Influencing the Response to Infection with SARS-COV-2
Brief Title: Genetic and Immunologic Basis of COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ali Sobh, Lecturer of Pediatric Immunology, Mansoura University
Other Study IDs: RP:20.05.70
Record Dates: First submitted 2020-05-10; First posted 2020-05-12 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Genetic Basis of COVID-19 Infection
Keywords: SARS-COV-2, Genetics
MeSH Terms: interventions — Exome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Whole Exome Sequencing — Genetic study of patients

SUMMARY:
We will study genetic factors causing severe disease due to infection with SARS-COV-2 which may help to find targeted therapy

ELIGIBILITY:
Inclusion Criteria:

* severe COVID-19 infection

Exclusion Criteria:

* Comorbidity ((DM, hypertension, Chronic liver or Kidney diseases, HIV, morbid obesity, Malignancy, Immunosuppressive therapy)

Ages: 1 Day to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: COVID-19 positive patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Mutations leading to increase susceptibility to SARS-COV-2 infection | 12 months
  Genetic susceptibility to COVID-19

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlyia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided